CLINICAL TRIAL: NCT05490316
Title: A Phase I Randomized, Double-Blind, Placebo-Controlled, Multiple Oral Dose Trial to Assess the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic of IBI353 (Orismilast) in Healthy Subjects
Brief Title: A Study of IBI353 (Orismilast) in Chinese Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI353A101
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo tablet (Placebo Comparator)
  Interventions: Drug: placebo
- IBI353 (Orismilast) dose 2 (Experimental)
  Interventions: Drug: IBI353 (Orismilast)
- IBI353 (Orismilast) dose 1 (Experimental)
  Interventions: Drug: IBI353 (Orismilast)

INTERVENTIONS:
Drug: IBI353 (Orismilast) — dose 1 or dose 2
  Arms: IBI353 (Orismilast) dose 1; IBI353 (Orismilast) dose 2
Drug: placebo — placebo
  Arms: Placebo tablet

SUMMARY:
This is a first in Chinese population study to evaluate the safety, tolerability, PK and PD of multiple dose of modified-release IBI353 administered orally in healthy subjects. The study enrolls 20 healthy subjects and consists of 1 week of screening, 3 weeks of treatment period and 1 week of safety follow up after completion of last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female 18 to 45 years of age at the time of consent
2. BMI of 19-27Kg/m2 and weight of 50-100kg (male) or 45-100kg (female)
3. Participants are in good health condition at screening stage based on past history, lab tests, EEG, physical examinations, and vital signs.
4. Must provide written informed consent, and in the investigator's opinion, subject is able to understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the protocol restrictions and requirements

Exclusion Criteria:

1. Subjects who have a medical history of liver, kidney, cardiovascular, nervous / mental, gastrointestinal, respiratory, urinary, endocrine system;
2. Subjects who have a history of relapse or chronic infection, or a history of acute infection treated by antibiotics within 3 months;
3. Subjects who have previously used PDE4 inhibitor dugs;
4. Subjects who have clinically significant abnormalities determined by vital signs, physical examination, and laboratory measurements;
5. Subjects who are not suitable for this trial due to other reasons In the investigator' opinion

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Time to Maximal Blood Concentration (Tmax) of IBI353 and its related metabolites. | Baseline through Day 21
Maximal Concentration (Cmax) of IBI353 and its related metabolites. | Baseline through Day 21
Area Under the Concentration Curve (AUC) of IBI353 and its related metabolites. | Baseline through Day 21
Volume of Distribution (Vd/F) of IBI353 and its related metabolites. | Baseline through Day 21
Half life time of IBI353 and its related metabolites. | Baseline through Day 21
Clearance (CL/F) of IBI353 and its related metabolites. | Baseline through Day 21
Accumulation Ratio of IBI353 and its related metabolites. | Baseline through Day 21

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), gastrointestinal AEs, and changes of vital signs, lab examinations, physical examinations, ECGs in healthy subjects after drug administration. | Baseline through Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No